CLINICAL TRIAL: NCT00023010
Title: Follow-Up of a Phase-I Gene Therapy Trial of Patients With Leukocyte Adherence Deficiency
Brief Title: Gene Therapy for Patients With Leukocyte Adherence Deficiency (Follow-Up of Phase 1 Trial)
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010236; 01-C-0236; NCT00004470 (obsolete NCT alias)
Record Dates: First submitted 2001-08-18; First posted 2001-08-20 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-12-13

CONDITIONS: Leukocyte Adhesion Deficiency Syndrome
Keywords: CD18; Retrovirus; RCR; Stem Cell; Gene Transfer; Leukocyte Adhesion Deficiency; LAD
MeSH Terms: conditions — Leukocyte-Adhesion Deficiency Syndrome; Leukocyte adhesion deficiency type 1

SUMMARY:
This study will provide long-term monitoring of two patients who received gene therapy for leukocyte adherence deficiency (LAD) under the Food and Drug Administration investigational new drug study BB-IND-7949. The IND protocol has been closed. No other patients are eligible for this study.

Patients previously enrolled in BB-IND-7949 (Retrovirus-Mediated Transfer of the cDNA for Human CD18 into Peripheral Blood Repopulating cells of Patients with Leukocyte Adherence Deficiency) will be followed at least yearly for an indefinite period of time to evaluate their medical status and look for treatment side effects. The follow-up visits at the NIH Clinical Center will involve the following:

* Interview regarding health status during the past year
* Blood draw of approximately 15 milliliters for 3 years, then 5 ml annually thereafter for studies related to LAD and to make sure no unexpected effects of gene therapy have occurred

The blood samples collected at the follow-up visits will be frozen and stored. If a serious medical problem arises, the sample may be checked for replication competent virus. If the gene therapy is suspected to be related to a medical problem, investigation may include a review of the patient's medical records or collection of additional blood or tissues for testing. If the patient should die, the family will be asked permission to perform an autopsy, regardless of the cause of death. Tissues taken at autopsy will be tested for any long-term effects from the gene therapy.

DETAILED DESCRIPTION:
Patients with leukocyte adhesion deficiency or LAD have a deficiency of the leukocyte integrin CD18 on their leukocyte cell surface and suffer from severe bacterial infections. Two patients with LAD were enrolled in a Phase I clinical trial conducted at the University of Washington School of Medicine in 1999 to determine the safety and potential efficacy of using retroviral vectors containing CD18 to transduce and correct their CD34+ peripheral blood stem cells. This protocol aims to continue the long-term follow-up of these patients at the National Cancer Institute where Dr. Hickstein is now a Senior Investigator. Blood samples will be collected at the follow-up visits on the yearly anniversary of the treatment date (either locally or off-site by the patients' personal physicians) for archiving for potential testing for replication competent retrovirus, and for complete blood counts. Patients will also undergo a history and physical examination at these visits. Results from these tests will be forwarded to the investigators who will report to the NIH and FDA.

ELIGIBILITY:
* Two patients treated under FDA IND BB-IND-7949.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2001-08-15; Study Completion 2010-12-13

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Anderson DC, Schmalsteig FC, Finegold MJ, Hughes BJ, Rothlein R, Miller LJ, Kohl S, Tosi MF, Jacobs RL, Waldrop TC, et al. The severe and moderate phenotypes of heritable Mac-1, LFA-1 deficiency: their quantitative definition and relation to leukocyte dysfunction and clinical features. J Infect Dis. 1985 Oct;152(4):668-89. doi: 10.1093/infdis/152.4.668. PMID 3900232
- [Background] Anderson DC, Springer TA. Leukocyte adhesion deficiency: an inherited defect in the Mac-1, LFA-1, and p150,95 glycoproteins. Annu Rev Med. 1987;38:175-94. doi: 10.1146/annurev.me.38.020187.001135. PMID 3555290